CLINICAL TRIAL: NCT01970033
Title: A Multicenter Randomized, Double-blind, Placebo Controlled ,Parallel Group ,Phase III Study to Access the Efficacy and Safety of SP2086 Treated Type 2 Diabetes Patients
Brief Title: Efficacy and Safety of SP2086 as Monotherapy in Patients With Type 2 Diabetes
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HR-SP2086-301
Record Dates: First submitted 2013-10-18; First posted 2013-10-25 (Estimated); Last update posted 2013-10-25 (Estimated); Status verified 2013-10

CONDITIONS: Type 2 Diabetes
Keywords: SP2086; Phase III; Monotherapy
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- SP2086 50 mg b.i.d (Experimental)
  Interventions: Drug: SP2086 50 mg b.i.d.
- SP2086 100 mg q.d. (Experimental)
  Interventions: Drug: SP2086 100 mg q.d.

INTERVENTIONS:
Drug: Placebo — * Run in period ：oral tablets of Placebo twice daily for 2 weeks
  * Phase A : oral tablets of Placebo twice daily for 24 weeks
  * Phase B : SP2086 50 mg b.i.d or SP2086 100 mg q.d. for 28 weeks
  Arms: Placebo
Drug: SP2086 50 mg b.i.d. — * Run-in period: placebo twice daily for 2 weeks
  * Phase A:SP2086 50 mg b.i.d for 24 weeks
  * Phase B:SP2086 50 mg b.i.d for 28 weeks
  Arms: SP2086 50 mg b.i.d
Drug: SP2086 100 mg q.d. — * Run-in period:placebo twice daily for 2 weeks
  * Phase A: SP2086 100 mg q.d. for 24 weeks
  * Phase B: SP2086 100 mg q.d. for 28 weeks
  Arms: SP2086 100 mg q.d.

SUMMARY:
SP2086 is a new dipeptidy1 peptidase(DPP)-4 inhibitors. This study aims to evaluate the efficacy and safety of SP2086 as monotherapy in patients with Type 2 Diabetes Mellitus in Metformin monotherapy Who Have Inadequate Glycemic Control treated with diet and exercise for 3 months

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with type 2 diabetes mellitus
* Patients have treated with diet/exercise at least 3 months
* 7.5% ≤HbA1C ≤11.0% at screening,7.0% ≤HbA1C ≤10.5% after run-in

Exclusion Criteria:

* Patient has history of type 1 diabetes mellitus
* Patient has history of ketoacidosis
* Patient has history of severe unconscious hypoglycemosis
* Patient has history of acute and chronic pancreatitis or pancreatic injury that may lead to high risk of pancreatitis
* Patient has history of decompensated heart failure (NYHA class III and IV), unstable angina, stroke or transient ischemic attack, myocardial infarction, persistence and clinical
* Patient has history of a history of hypertension, and after antihypertensive treatment, systolic blood pressure ≥ 160 mmHg or diastolic blood pressure ≥ 100 mmHg
* Patient has severe liver or kidney disease,alanine aminotransferase >2×UNL, Aspartate Aminotransferase >2×upper normal limit(UNL)；total bilirubin >2×UNL； creatinine>1.5 mg/dL (Male,132.6μmol/L) ，>1.4 mg/dL(Female，123.8μmol/L)
* Patient has severe chronic gastrointestinal disease or therapy that may affect drug absorption, such as gastrointestinal surgery
* Patient has severe haematological diseases or other diseases leading to hemolyze and red blood cell unstable (malaria、haemolytic anaemia eg. )
* Patient has other endocrine diseases, for example hyperthyroidism、hypothyroidism、hypercortisolism、multiple endocrine neoplasia and so on
* Patient has history of malignancy
* Patient has history of alcohol or drug abuse

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 450 (Estimated)
Dates: Start 2012-12; Primary Completion 2014-01 (Estimated); Study Completion 2015-01 (Estimated)

PRIMARY OUTCOMES:
Change From Baseline in HbA1c (Hemoglobin A1C) at Week24 | baseline, week 24
  A1C is measured as a percent. Thus, this change from baseline reflects the Week 24 A1C percent minus the Week 0 A1C percent

SECONDARY OUTCOMES:
Change From Baseline in fasting plasma glucose (FPG) at Week 24 | Weeks 0-24
  Change from baseline at Week 24 is defined as Week 24 FPG minus Week 0 FPG
Change From Baseline in 2-hour Post-meal Glucose (2-hr PMG) at Week 24 | Weeks 0-24
  Change from baseline at Week 24 is defined as Week 24 2-hr PMG minus Week 0 2-hr PMG
Percentage of Participants Achieving Less Than (<) 6.5% or <7% HbA1c Levels | week24
Change From Baseline in A1C at Week 52 | week 52
  A1C is measured as a percent. Thus, this change from baseline reflects the Week 52 A1C percent minus the Week 0 A1C percent
Change From Baseline in FPG at Week 52 | week 52
  Change from baseline at Week 52 is defined as Week 104 FPG minus Week 0 FPG
Change From Baseline in lipid at Week 4、8、12、24、38、52 | Week 4、8、12、24、38、52
Change From Baseline in Body Weight at Week 4,8,12、24、38、52 | Week 4、8、12、24、38、52

CONTACTS AND LOCATIONS:
Overall Officials: Changyu Pan, M.D., Principal Investigator — Chinese PLA General Hospital
Locations (1):
- Chinese PLA General Hospital, Beijing, China